CLINICAL TRIAL: NCT06743074
Title: Effectiveness of Different Exercise Programmes in Individuals With Dynamic Knee Valgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: hazal genc (Other)
Responsible Party: Sponsor-Investigator, hazal genc, Principal Investigato, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: e-10840098
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Knee Valgus
Keywords: knee; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- foot Exercise (Experimental): foot exercise
  Interventions: Other: foot exercise
- hip exercise (Experimental): hip exercise
  Interventions: Other: hip exercise
- control group (Other): other
  Interventions: Other: control

INTERVENTIONS:
Other: foot exercise — foot exercise
  Arms: foot Exercise
Other: hip exercise — hip exercise
  Arms: hip exercise
Other: control — control
  Arms: control group

SUMMARY:
Dynamic knee valgus (DDV) is an erroneous movement pattern of the lower limb that occurs in multiple planes. It results from a combination of hip joint adduction, femoral anteversion, knee abduction and external tibial torsion .

DETAILED DESCRIPTION:
Dynamic knee valgus (DDV) is an erroneous movement pattern of the lower limb that occurs in multiple planes. It results from a combination of hip joint adduction, femoral anteversion, knee abduction and external tibial torsion . DDV is also referred to as a mechanism in which the knee joint moves medially relative to the hip and foot with the centre fixed to the ground.

ELIGIBILITY:
Inclusion criteria:

* Age between 18-50 years.
* Absence of any lower extremity pain.
* Having a frontal plane projection angle of 10 and above in the descent phase of squatting on one leg.
* Having active or regular physical activity.
* Volunteering to participate in the study.

Exclusion criteria:

* Active knee pain.
* History of patellar instability.
* Presence of rheumatic diseases such as osteoarthritis, rheumatoid arthritis.
* History of trauma or injury causing ligament laxity in the ankle, hip or knee.
* Having a neurological disease that may impair the ability to perform any lower limb movement.
* Having undergone any lower extremity surgery before.
* Having received physiotherapy from hip, knee and ankle in the last 6 months.
* To be benefiting from another treatment during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Frontal Plane Projection Angle (FPPA) | 6 weeks
  FPPA is measured as the angle between a line drawn from the marked point on the proximal thigh to the knee joint and another line extending from the knee joint to the ankle during maximum knee flexion. A 2D analysis is performed through single-leg squat (SLS), vertical jump (VJ), and single-leg landing (SLL). An increase of 10° or more in FPPA during a single-leg squat is categorized as "Observable Dynamic Knee Valgus (DKV)."
Lower Extremity Clinical Measurements | 6 weeks
  Clinical measurements help assess the functional performance of the lower extremities and prevent injuries. Key parameters include Q-angle, hip anteversion angle, tibial torsion, ankle dorsiflexion, and rearfoot angle. Standardized tests such as goniometer-based Q-angle measurement, Craig's test for hip anteversion, and subtalar joint neutral positioning for dorsiflexion are utilized.
Balance Evaluation | 6 weeks
  Static balance was assessed with the Single Leg Stance Test (SLST), while dynamic balance was evaluated using the Y Balance Test (YBT) in three directions: anterior, posteromedial, and posterolateral.
Proprioception Assessment | 6 weeks
  Proprioception was evaluated using the Active Joint Position Sense (AJPS) test, which measures the ability to replicate a target angle. Measurements were conducted with a Baseline digital goniometer, and angular deviation was recorded to determine accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: aleyna zeynep karcıoğlu, Study Chair — Bahçeşehir University
Locations (1):
- bahcesehır University, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No